CLINICAL TRIAL: NCT03191578
Title: A Randomized, Double-Blind, Placebo-Controlled Phase I Trial to Evaluate the Immunomodulatory Effect of RUTI® in Individuals With High-Risk Non-Muscle-Invasive Bladder Cancer (NMIBC) Treated With Intravesical Bacillus Calmette-Guerin (BCG)
Brief Title: Immunological Response to Intravesical BCG Therapy of Superficial Bladder Cancer by Prior Administration of RUTI®
Acronym: RUTIVAC-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Archivel Farma S.L. (Industry)
Collaborators: Fundació Institut Germans Trias i Pujol (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: RUTIVAC-1
Record Dates: First submitted 2017-06-09; First posted 2017-06-19 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: High-Risk Non-Muscle-Invasive Bladder Cancer
Keywords: NMIBC; Immunotherapy; RUTI; Non-muscle invasive bladder cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RUTI® injection (Experimental)
  Interventions: Drug: RUTI®
- Sodium Chloride 0.9% injection (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RUTI® — Administration of RUTI®
  Arms: RUTI® injection
Drug: Placebo — Administration of placebo
  Arms: Sodium Chloride 0.9% injection

SUMMARY:
The RUTIVAC-1 study is a Phase I Clinical Trial designed to evaluate the systemic and mucosal immunological response and provide safety information after the use of RUTI® administration to individuals with NMIBC.

The study will enroll individuals treated with Transurethral resection of bladder tumor (TURBT), diagnosed to have high-risk Non-muscle invasive bladder cancer (NMIBC) and suitable candidates for BCG therapy and who meet all eligibility criteria.

Forty individuals will be recruited and randomized 1:1 to receive two subcutaneous shots of 25 μg RUTI® or placebo. After vaccination, individuals will receive the standard induction course, of intravesical Bacillus Calmette-Guerin (BCG)therapy (weekly BCG for six weeks).

4 to 8 weeks after the last intravesical BCG administration (BCG6) a visit will be performed (Visit 1, end of the interventional phase). Once all participants have performed VISIT 1 immunological assays will be performed and data will be analyzed.

At the end of the Interventional Phase the blind will be opened, except for the study physicians who will remain blind during all the follow-up. All the individuals will be followed up for three years since TURBT.

ELIGIBILITY:
Inclusion Criteria:

1. Written ICF for participation in the study.
2. Age ≥18 years.
3. General health status according to WHO ≤ 2.
4. Have primary histologically confirmed T1 and/or high grade tumors and/or CIS.
5. All visible papillary tumors must be completely resected.
6. Early postoperative (within 24 hours of TURBT) single dose chemotherapy is allowed.
7. BCG therapy indication.
8. Never treated with BCG immunotherapy
9. Willing to comply with study visits and procedures as per protocol
10. Use of reliable contraception (see section 8.6) from the screening visit to 30 days after the last RUTI® or placebo injection.

Exclusion Criteria:

1. Life expectancy <5 years.
2. Have a severe concomitant disease that might limit compliance or completion of the protocol.
3. Have any other malignancy that might impact 3-year survival or might be potentially confused with NMIBC.
4. Have other neoplasms.
5. Have congenital or acquired immune deficiencies or under immunomodulatory treatment.
6. Be receiving cytotoxic drugs or systemic corticosteroids within 8 weeks of receiving the first administration of BCG.
7. Have received radiation therapy for their bladder cancer within 4 months prior to study entry.
8. Have active infections (including urinary tract infections) defined as viral, bacterial, or fungal infections requiring therapy, HIV-positive status, concurrent febrile illness, gross hematuria or other factor that could influence tolerability to intravesical BCG therapy.
9. Have biopsy, TURBT, or traumatic catheterization within 14 days of start of intravesical BCG treatment.
10. Have active tuberculosis at screening visit.
11. Active pregnancy or breastfeeding.
12. Soy allergy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Changes in the systemic Th1 immune response. | Baseline, Day 10, weeks 2, 7 and 16
  IFN-γ production assessed by intracellular staining after ex vivo stimulation of PBMCs with PPD
Changes in the local immune response in peritumoral tissue (Th1/Th2 ratio) | Baseline and week 16 visit
  Th1/Th2 ratio in cells in the peritumoral tissue
Changes in the local immune response in urine | Baseline, Day 10, weeks 2, 7 and 16
  Urine levels of cytokines by multiplex analysis

SECONDARY OUTCOMES:
Recurrence date | Until 3 years since TURBT
  Recurrence date
Disease worsening | Until 3 years since TURBT
  Disease worsening: events that included diagnosis of T2 or greater
Death | Until 3 years since TURBT
Proportion of patients who develop a Grade 3 or 4 local reactions | through study completion an average of 1,5 year
  From Baseline to BCG administration number 6
Proportion of patients who develop a Grade 3 or 4 systemic reactions | through study completion an average of 1,5 year
  Proportion of patients who develop a Grade 3 or 4 systemic reactions (adverse events related to RUTI/placebo).

CONTACTS AND LOCATIONS:
Locations (1):
- Germans Trias i Pujol Hospital, Badalona, Barcelona, Spain